CLINICAL TRIAL: NCT01060774
Title: Comparison of Bupivacaine vs Lidocaine on Inflammatory Regulation Following Endodontic Surgery: A Double-Blind, Randomized, Controlled Clinical Trial
Brief Title: Bupivacaine Versus Lidocaine on Inflammatory Regulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland (Other)
Responsible Party: Principal Investigator, Sharon Gordon, Associate Professor, University of Maryland
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HP-00043039
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Pain
Keywords: Bupivacaine; Inflammation; Pain; Local Anesthetic; peripheral sensitization
MeSH Terms: conditions — Pain; Inflammation | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Experimental): 0.5% bupivacaine/1:200,000 epinephrine
  Interventions: Drug: Bupivacaine
- Lidocaine (Experimental): 2% lidocaine/1:200,000 epinephrine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Up to 5 capsules of 2% lidocaine with epinephrine as a reinforcement drug post-operatively
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Bupivacaine — Up to 5 capsules of 0.5% Bupivacaine with epinephrine given post-operatively.
  Other Names: Marcain, Marcaine, Sensorcaine and Vivacaine.
  Arms: Bupivacaine

SUMMARY:
This study is testing a local anesthetic (numbing medicine) to suppress pain. Bupivacaine and lidocaine are FDA approved local anesthetics that may decrease pain following surgery. Patients will receive either 2% lidocaine, 0.5% bupivacaine, or placebo with epinephrine 1:200,000 as a numbing medicine at the end of root canal surgery. Small pieces of gum will be taken before and after surgery and 2 days later to analyze chemicals that may be related to pain sensation.

DETAILED DESCRIPTION:
We hypothesize that the use of the LLA bupivacaine will promote local inflammation leading to increased pain and central sensitization as evaluated by increase in pain at later time points. Hence our main hypothesis to be evaluated and statistically tested for our primary endpoint (Aim 1) is:

HO: There is no difference in mean levels of biochemical mediators of inflammation between groups.

HA: The bupivacaine group has higher levels of biochemical mediators following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers referred for endodontic surgery willing to undergo 2 visits: 1 surgical appointment, and 1 follow-up research-related appointment
* Ages of 18 and older
* Willing to undergo observation for 1/2 hour post-operatively
* Willing to complete a 100 mm visual analog scale and record analgesic intake over 48 hrs period
* Willing to have a preoperative and postoperative biopsy on the day of surgery
* Willing to return at 48 hours post-operation to turn in completed pain diaries and for the third biopsy

Exclusion Criteria:

* Allergy to or other contraindications to use of aspirin, sulfites, amide anesthetics, or acetaminophen
* Chronic use of medications confounding the assessment of the inflammatory response or analgesia, for example, NSAIDS, COX-2 inhibitors, antihistamines, steroids, antidepressants
* Medications contraindicated with bupivacaine: MAO inhibitors and anti-depressants
* Diseases such as diabetes mellitus, liver disease, chronic infections, rheumatoid arthritis or any other systemic disease that compromises the immune system
* Unusual surgical difficulty

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Assess the local inflammatory response as measured by tissue expression of the prostanoid enzymes cyclooxygenase (COX-2) and other cytokines and inflammatory mediators. | 48 hours
  The difference in inflammatory gene expression between treatment groups.

SECONDARY OUTCOMES:
Evaluate the clinical outcome of postoperative pain following endodontic surgery, as measured by pain category and visual analog scale (VAS) and postoperative analgesic requirements. | 48 hours
  The subject-reported pain measured at 48 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Gordon, Principal Investigator — University of Maryland, Baltimore College of Dental Surgery; Anastasia Mischenko, Study Director — University of Maryland, Baltimore College of Dental Surgery; Morris Hicks, Study Director — University of Maryland, Baltimore College of Dental Surgery; Ashraf Fouad, Study Director — University of Maryland, Baltimore College of Dental Surgery
Locations (1):
- University of Maryland, Baltimore College of Dental Surgery, Baltimore, Maryland, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT01060774/Prot_SAP_000.pdf